CLINICAL TRIAL: NCT07033572
Title: Hybrid Endoscopic Hemithyroidectomy and Targeted Ablation for Bilateral Papillary Thyroid Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Director, Head of Thyroid Surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hybrid
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Thyroid Neoplasms; Carcinoma, Papillary
Keywords: Hybrid endoscopic thyroidectomy; Radiofrequency ablation; Thyroid function preservation; Bilateral Thyroid Carcinoma
MeSH Terms: conditions — Thyroid Neoplasms; Carcinoma, Papillary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid Endoscopic Hemithyroidectomy + Same-Session Contralateral RFA (Experimental): Remote-access gas-less axillo-breast endoscopic hemithyroidectomy with level VI central-neck dissection on the dominant lobe, immediately followed-under the same anesthesia-by ultrasound-guided radiofrequency ablation (17-G, 0.7 cm active tip, 40 W, moving-shot technique) of a ≤ 7 mm contralateral papillary thyroid microcarcinoma.
  Interventions: Procedure: Endoscopic Hemithyroidectomy with Central-Neck Dissection; Procedure: Ultrasound-Guided Radiofrequency Ablation of Contralateral Nodule

INTERVENTIONS:
Procedure: Endoscopic Hemithyroidectomy with Central-Neck Dissection — Gas-less axillo-breast approach (trans-axillary + peri-areolar), carbon-dioxide-free working space, removing dominant thyroid lobe plus level VI lymph nodes; intra-operative neuromonitoring used throughout.
Procedure: Ultrasound-Guided Radiofrequency Ablation of Contralateral Nodule — 17-gauge internally-cooled electrode, 0.7 cm active tip, power 40 W; moving-shot technique under real-time ultrasound until hyperechoic halo fully covers ≤ 7 mm papillary microcarcinoma ≥ 2 mm from posterior capsule; same anesthesia session as surgery.

SUMMARY:
This study evaluates a thyroid-function-preserving alternative to routine total thyroidectomy for bilateral papillary thyroid carcinoma (PTC). Eligible adults undergo remote-access gas-less axillo-breast endoscopic hemithyroidectomy with level VI dissection on the dominant side, followed by ultrasound-guided radiofrequency ablation (RFA) of a ≤7 mm contralateral focus during the same anesthesia. Outcomes include structural-recurrence-free survival, endocrine-function preservation, safety, and quality of life over 24 months.

DETAILED DESCRIPTION:
Bilateral PTC traditionally prompts total thyroidectomy, exposing patients to lifelong thyroxine replacement and a 1 - 3 % risk of permanent hypocalcemia. Building on a pilot cohort of 11 patients treated from June 2018 to September 2024 that showed no structural recurrence, no permanent RLN palsy, and preserved endocrine function after a median 17-month follow-updraft_Proof_hi, we launch a multicenter registry to confirm oncologic adequacy and functional benefits. Intervention: endoscopic hemithyroidectomy (dominant lobe) via gas-less axillo-breast approach plus central-neck dissection; then contralateral lesion RFA with a 17-gauge 0.7-cm active-tip electrode at 40 W (moving-shot). Follow-up at 1, 6, 12, 18, and 24 months includes ultrasound, serum Tg, calcium, PTH, and QoL instruments. Long-term surveillance continues annually to five years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Dominant-side PTC ≤1.5 cm suitable for endoscopic resection.
* Contralateral nodule ≤7 mm located ≥2 mm from posterior capsule.
* No radiologic lymph-node metastasis on contralateral side.
* Written informed consent.

Exclusion Criteria:

* Extrathyroidal extension, gross nodal or distant metastasis.
* Prior neck surgery, prior RFA/ethanol injection, or neck irradiation.
* Pregnancy or lactation.
* Serious comorbidities precluding anesthesia or follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Structural Recurrence-Free Survival | 24 months
  Proportion of participants without local, regional, or distant structural recurrence confirmed by imaging ± cytopathology.
Endocrine-Function Preservation | 24 months
  Participants alive and free from lifelong levothyroxine therapy and permanent hypocalcemia (serum Ca ≥2.1 mmol/L without supplementation).

SECONDARY OUTCOMES:
Permanent RLN Palsy Incidence | 12 months
  Laryngoscopy-confirmed vocal-fold mobility disorder persisting ≥6 months.
Permanent Hypocalcemia Incidence | 12 months
  Need for calcium/vit-D >6 months after surgery.
Nodule Volume Reduction Rate | 12 months
  Percentage reduction of ablated nodule volume on ultrasound.
Procedure-Related Adverse Events | 30 days
  Any CTCAE v5.0 Grade ≥3 event within 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang MD, Principal Investigator, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No